CLINICAL TRIAL: NCT05420675
Title: Vastus Medialis Muscle Activation During Single Leg Squat Performed With Arm Position Variations in Healthy Participants
Brief Title: Different Arm Positions During Single Leg Squat
Status: Completed | Type: Observational
Sponsor: Hacettepe University (Other)
Responsible Party: Principal Investigator, Gökhan Karakaş, Principal Investigator, Hacettepe University
Other Study IDs: GO22-582
Record Dates: First submitted 2022-06-11; First posted 2022-06-15 (Actual); Last update posted 2022-09-02 (Actual); Status verified 2022-08

CONDITIONS: Knee Injuries and Disorders
Keywords: healthy subject; movement analysis; muscle activity; kneeling
MeSH Terms: conditions — Knee Injuries; Disease

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Single Leg Squat — After initial data collection (Demographic data, Inclusion criteria), surface electromyography EMG assessments will be obtained from 1 muscle ( Vastus Medialis). EMG evaluation will be done in different arm positions during the single leg squat. These records will be taken in 4 different situations: 1) Arms free, 2) Arms flexed to 90 degrees, 3) Hands on hips, 4) Arms across the chest.

SUMMARY:
The aim of this study is to compare the effects of different arm positions on muscle activity during single leg squat.

DETAILED DESCRIPTION:
The aim of our study is to examine the effect of different positions of the arms on lower extremity muscle activations during Single Leg Squat (SLS). This prospective cross sectional study included single leg squat test assessments in different arm positions: 1) Arms free, 2) Arms flexed 90 degrees, 3) Hands on hip, 4) Arms across the chest. Inclusion criteria were being a young adult (20-30 years old), physical activity level of at least 4 on the Tegner Activity Scale, and volunteering to participate in the study. Those with a history of lower extremity injury in the last 1 year will be excluded from the study. Our study will contribute to distinguishing SLS variations for clinicians and researchers and choosing the appropriate SLS for evaluation and treatment.

ELIGIBILITY:
Inclusion Criteria:

* Being between the ages of 20-30
* Physical activity level of at least 4 on the Tegner Activity Scale,

Exclusion Criteria:

* History of lower extremity injury in the last 1 year
* Central or peripheral vestibular disorders

Ages: 20 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Healthy Volunteers
Sampling Method: Probability Sample
Enrollment: 20 (Actual)
Dates: Start 2022-06-08 (Actual); Primary Completion 2022-07-15 (Actual); Study Completion 2022-08-01 (Actual)

PRIMARY OUTCOMES:
Surface Electromyography | Procedure (During the intervention)
  Surface EMG evaluations of Vastus Medialis in 4 conditions in a row (1) Arms free, 2) Arms flexed 90 degrees, 3) Hands on hip, 4) Arms on crossed shoulders.

CONTACTS AND LOCATIONS:
Overall Officials: Gözde Yağcı, Assoc.Prof., Study Director — Hacettepe University Faculty of Physical Therapy and Rehabilitation; Semra Topuz, Prof., Principal Investigator — Hacettepe University Faculty of Physical Therapy and Rehabilitation; Gökhan Karakaş, M.Sc., Principal Investigator — Hacettepe University Faculty of Physical Therapy and Rehabilitation; Alev Doğan, M.Sc., Principal Investigator — Hacettepe University Faculty of Physical Therapy and Rehabilitation; Ali Yalçın, M.Sc., Principal Investigator — Hacettepe University Faculty of Physical Therapy and Rehabilitation
Locations (1):
- Hacettepe University, Faculty of Physical Therapy and Rehabilitation, Department of Physiotherapy and Rehabilitation, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided